CLINICAL TRIAL: NCT02413424
Title: Metabolic Effects of Non-nutritive Sweeteners
Acronym: NNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 201412080; P30DK020579 (NIH)
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Obesity
Keywords: sucralose
MeSH Terms: conditions — Obesity | interventions — trichlorosucrose; Water

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Drink Sucralose (Experimental): Subjects will drink sucralose 10 min before drinking a glucose load
  Interventions: Dietary Supplement: Sucralose; Dietary Supplement: glucose load
- Drink Water (Placebo Comparator): Subjects will drink water 10 min before drinking a glucose load
  Interventions: Other: Water; Dietary Supplement: glucose load
- Taste and spit Sucralose (Experimental): Subjects will taste and spit up sucralose 10 min before drinking a glucose load
  Interventions: Dietary Supplement: Sucralose; Dietary Supplement: glucose load

INTERVENTIONS:
Dietary Supplement: Sucralose — 60 ml of 2mM sucralose
  Arms: Drink Sucralose; Taste and spit Sucralose
Other: Water — 60 ml of water
  Arms: Drink Water
Dietary Supplement: glucose load

SUMMARY:
The purpose of this research study is to examine whether sugar-replacement sweeteners that are currently on the market (ex. Sucralose, which is in Splenda) change how well the body works to control blood sugar.

DETAILED DESCRIPTION:
The investigators of this study have recently found that sucralose, the most commonly used non-nutritive sweetener (NNS), affects the glycemic response to an oral glucose tolerance test (OGTT) and potentiates glucose-stimulated insulin secretion in obese people who are not regular consumers of NNS. However, studies conducted in healthy lean adults, none of which control for previous use of NNS, show that sucralose does not affect glycemic or hormonal responses to the ingestion of glucose or other carbohydrates. Therefore, we do not know a) whether sucralose effects are limited to obese subjects, or are generalizable to lean people when controlling for prior history of NNS consumption, and b) mechanism(s) responsible for the acute effect of sucralose on glucose metabolism as we measured in obese subjects. The aim of this study is to determine the effects of an acute intake of sucralose on the metabolic response to an oral glucose tolerance test in lean and obese people.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 kg/m2 or BMI ≥ 18 kg/m2 and BMI<25 kg/m2
* "insulin sensitive": based on the homeostasis model assessment of insulin resistance (HOMA-IR) <3

Exclusion Criteria:

* BMI ≥ 25 kg/m2 and BMI<30 kg/m2
* HOMA-IR>3
* Current smoker or quit smoking less than 6 months ago
* pregnancy or breastfeeding
* subjects who have malabsorptive syndromes, phenylketonuria, inflammatory intestinal disease, liver or kidney diseases, diabetes
* subjects who are taking any medication that might affect metabolism
* anemia
* regular use of non-nutritive sweeteners

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Peak insulin secretion rate | up to 5 hours after drinking a glucose load
  Blood samples will be collected before and for 5 hours after drinking a glucose load to determine plasma insulin and C-peptide. Insulin secretion rate will be assessed using the minimal model of Breda and collaborators.
Glucose rate of appearance | up to 5 hours after drinking a glucose load
  Blood samples will be collected before and for 5 hours after drinking a glucose load to determine glucose and glucose tracer:tracee ratios.

SECONDARY OUTCOMES:
Glucose-dependent insulinotropic polypeptide (GIP) | up to 5 hours after drinking a glucose load
  Blood samples will be collected before and for 5 hours after drinking a glucose load to determine GIP.
Sucralose concentrations in plasma | up to 310 min after drinking the sucralose load
  Sucralose concentrations in plasma will be measured by using liquid chromatography-mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Y Pepino, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana Champaign, Urbana, Illinois, United States

REFERENCES:
- [Background] Pepino MY, Tiemann CD, Patterson BW, Wice BM, Klein S. Sucralose affects glycemic and hormonal responses to an oral glucose load. Diabetes Care. 2013 Sep;36(9):2530-5. doi: 10.2337/dc12-2221. Epub 2013 Apr 30. PMID 23633524
- [Background] Brown RJ, de Banate MA, Rother KI. Artificial sweeteners: a systematic review of metabolic effects in youth. Int J Pediatr Obes. 2010 Aug;5(4):305-12. doi: 10.3109/17477160903497027. PMID 20078374
- [Background] Margolskee RF, Dyer J, Kokrashvili Z, Salmon KS, Ilegems E, Daly K, Maillet EL, Ninomiya Y, Mosinger B, Shirazi-Beechey SP. T1R3 and gustducin in gut sense sugars to regulate expression of Na+-glucose cotransporter 1. Proc Natl Acad Sci U S A. 2007 Sep 18;104(38):15075-80. doi: 10.1073/pnas.0706678104. Epub 2007 Aug 27. PMID 17724332
- [Background] Swithers SE. Artificial sweeteners produce the counterintuitive effect of inducing metabolic derangements. Trends Endocrinol Metab. 2013 Sep;24(9):431-41. doi: 10.1016/j.tem.2013.05.005. Epub 2013 Jul 10. PMID 23850261
- [Background] Suez J, Korem T, Zeevi D, Zilberman-Schapira G, Thaiss CA, Maza O, Israeli D, Zmora N, Gilad S, Weinberger A, Kuperman Y, Harmelin A, Kolodkin-Gal I, Shapiro H, Halpern Z, Segal E, Elinav E. Artificial sweeteners induce glucose intolerance by altering the gut microbiota. Nature. 2014 Oct 9;514(7521):181-6. doi: 10.1038/nature13793. Epub 2014 Sep 17. PMID 25231862